CLINICAL TRIAL: NCT03592108
Title: Benefit of Cheyne-Stokes Respiration Remote Monitoring in CPAP-treated Patients With Obstructive Sleep Apnea for the Early Detection of Significant Cardiac Events.
Brief Title: Benefit of Cheyne-Stokes Respiration Remote Monitoring in CPAP-treated Patients With Obstructive Sleep Apnea to Detect Early Events of Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Medical de Pneumologie, Polyclinique Saint-Laurent (Other)
Collaborators: Slb Pharma (Other); VitalAire (Industry); Regional Health Agency - Brittany (Other); ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AlertApnée
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea (OAS); Cheyne-Stokes respiration (CSR); Continuous positive airway pressure (CPAP); Telemedicine; Heart failure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cheyne-Stokes Respiration; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CSR remote monitoring (Experimental): The remote monitoring of CPAP treatment will be modified in order to detect the presence of CSR as soon as any significant increase of the apnea-hypopnea index occurs.
  Interventions: Other: CSR remote monitoring

INTERVENTIONS:
Other: CSR remote monitoring — The intervention will consist to modify the method used to analyse the data collected by remote monitoring in OSA-patients treated by CPAP (device : AirSense™10 Autoset™, ResMed) in order to alert physicians when Cheynes-Stokes respiration (CSR) occurs during sleep and then to set up emergency pulmonology and cardiology consultations to screen the onset of a significant cardiac event (heart failure, rhythm disorder, diastolic dysfunction).

SUMMARY:
Obstructive sleep apnea (OSA) syndrome affects 40-60% of patients presenting with cardiovascular diseases. Cheyne-Stokes respiration is a type of central apnea characterised by the presence of at least three consecutive episodes of apnea and/or hypopnea separated by a crescendo-decrescendo variation of the breathing amplitude with a cycle length ≥ 40 seconds and a central apnea/hypopnea index ≥ 5/h, for at least two hours of recording.

The association between heart failure and Cheynes-Stokes respiration is known and a recent study showed that Cheynes-Stokes respiration was associated with more severe heart failure. Moreover, a medical and medical/financial benefit of the early detection of cardiac decompensation has been reported.

The purpose of this feasibility study is to investigate the benefit of Cheyne-Stokes respiration remote monitoring in CPAP-treated patients with OSA for the early detection of significant cardiac events (heart failure, rhythm disorder, diastolic dysfunction).

To achieve this aim, a modified approach of CPAP remote monitoring is proposed based on the performance of the latest generation of positive pressure devices from ResMed, AirSense™ 10 Autoset™, which can detect and record the presence of Cheynes-Stokes respiration. For a period of 12 months, in addition to the usual daily remote monitoring (CPAP adherence, pressure settings, level of air leakages), the healthcare provider will systematically monitor the CSR data whenever the AHI increases significantly. Physicians will be alerted when a CSR occurs and they will see the patients within a short time for pulmology and cardiology consultations in order to screen the onset of significant cardiac event.

After the 12-month period of modified remote monitoring, the telemedicine returns to the usual procedure. Patients who had at least one CSR occurrence during the first 12-month period will be followed up to 24 months to assess their medical condition.

ELIGIBILITY:
Inclusion Criteria:

* patient with severe OSA treated with CPAP (device AirSense™10 Autoset™ by ResMed).
* patient followed up by one of the lung specialist of the Polyclinique Saint-Laurent and tele-monitored by the healthcare provider VitalAire.

Exclusion Criteria:

* enrolled in an interventionnal clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Proportion of significant cardiac events following the detection of Cheyne-Stokes Respiration during sleep | 12 months
  To determine the correlation between the occurrence of Cheyne-Stokes Respiration during sleep and the onset of a significant cardiac event during the 12 month period of modified remote monitoring.

SECONDARY OUTCOMES:
Characterisation of apnea-hypopnea index and CPAP treatment when the Cheyne-Stokes Respiration occurs | throughout the 12 month period
  Each time a CSR is detected during sleep, the mean AHI of the last 7 days and the machine settings (the 95th percentile pressure, fixed or autoset mode, level of air leakages, other settings) will be monitored.

OTHER OUTCOMES:
CPAP treatment adherence | 12 months
  The mean number of nights with CPAP use > 4 hours
Medical condition of patients after CSR occurence | 24 months
  To assess the medical condition of patients who had at least one Cheyne-Stokes Respiration during the 12 months modified remote monitoring. The number of pulmonology and cardiology consultations and/or hospitalisations will be monitored up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Prigent, MD, Principal Investigator — Groupe Médical Pneumologie - Polyclinique Saint-Laurent
Locations (1):
- Polyclinique Saint-Laurent, Rennes, France

REFERENCES:
- [Derived] Prigent A, Pellen C, Texereau J, Bailly S, Coquerel N, Gervais R, Liegaux JM, Luraine R, Renaud JC, Serandour AL, Pepin JL. CPAP telemonitoring can track Cheyne-Stokes respiration and detect serious cardiac events: The AlertApnee Study. Respirology. 2022 Feb;27(2):161-169. doi: 10.1111/resp.14192. Epub 2021 Dec 6. PMID 34873795